CLINICAL TRIAL: NCT07046182
Title: Clinical Study of CEP+Dasatinib + Azacytidine in First-line Treatment of. Angioimmunoblastoma Foresight
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Zhengzhou University (Other)
Responsible Party: Principal Investigator, Mingzhi Zhang, professor, Zhengzhou University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-IIT-ZMZ/YJQ
Record Dates: First submitted 2025-06-22; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Angioimmunoblastic T-cell Lymphoma (AITL)
MeSH Terms: conditions — Immunoblastic Lymphadenopathy | interventions — Dasatinib; Azacitidine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- group1 (Experimental): CEP + Dasatinib + Azacitidine
  Interventions: Biological: CEP + Dasatinib + Azacitidine

INTERVENTIONS:
Biological: CEP + Dasatinib + Azacitidine — CEP + Dasatinib + Azacitidine as the first-line treatment regimen for patients with Angioimmunoblastic T-cell Lymphoma

SUMMARY:
To observe the efficacy and safety of the CEP + Dasatinib + Azacitidine as the first-line treatment regimen for patients with Angioimmunoblastic T-cell Lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* 1.Age 18-75 years, ECOG 0-2. 2.Life expectancy >6 months. 3.Pathologically confirmed AITL. 4.Acceptable hematological parameters (neutrophils ≥1.0×10⁹/L, platelets ≥75×10⁹/L, hemoglobin ≥80 g/L [except for bone marrow infiltration]).

  5.At least one measurable lesion (lymph node: long diameter ≥1.5 cm, short diameter ≥1.0 cm; extranodal: long diameter ≥1.0 cm).

  6.Liver function: TBIL ≤1.5×ULN, ALT/AST ≤2.5×ULN, ALP ≤3×ULN (non-bone infiltration).

  7.Renal function: serum creatinine ≤1.5×ULN. 8.No severe comorbidities; normal cardiac function. 9.Willingness to use contraception; negative pregnancy test for育龄期女性 (within 7 days prior to first dose).

  10.Informed consent and compliance with follow-up. 11.No concurrent anti-tumor therapies (e.g., traditional Chinese medicine, immunotherapy, biological agents).

Exclusion Criteria:

- 1.Patients with definite neurological or psychiatric diseases, including dementia or epilepsy, with a history of psychotropic drug abuse and inability to quit, or other substantive lesions that may increase central neurotoxicity; 2.Those who are participating in other clinical trials or have participated in other clinical research within the previous 4 weeks (except those who have not received treatment); 3.Systemic autoimmune diseases or immunodeficiency; 4.Refusal to provide blood samples; 5.Allergic to any drug in the plan; 6.Pregnant and lactating women; 7.Subjects with significant diseases that may interfere with the trial and with uncontrolled active infections; 8.Primary or relapsed central nervous system tumors; 9.Contraindications for chemotherapy; 10.Researchers believe that they are not suitable for inclusion; 11.Any active bacterial, viral, fungal, mycobacterial, parasitic or other infections (excluding superficial skin or mucosal infections) or any major systemic infectious diseases (septicemia, etc.) that require antibiotic treatment or hospitalization within the previous 4 weeks before inclusion; 12.Those who have received anti - tumor treatment (such as radiotherapy, chemotherapy, immunotherapy, biotherapy, immunotherapy); 13.Other severe conditions that may prevent the subject from participating in this trial, such as uncontrolled diabetes: Severe cardiac insufficiency (NYHA grade III or above); Acute coronary syndrome occurred within the previous 6 months; Coronary artery bypass grafting or stent implantation, mitral valve surgery, and other heart and major vascular - related surgeries within the previous 6 months; Severe arrhythmias including bradycardia, tachycardia, fast atrial fibrillation, atrial flutter, uncontrolled severe hypertension (systolic pressure ≥ 180 mmHg, diastolic pressure ≥ 110 mmHg), peptic ulcer disease (subjects judged to have a perforated peptic ulcer); Active autoimmune diseases (such as systemic lupus erythematosus, rheumatoid arthritis, polymyositis, scleroderma, autoimmune hemolytic anemia, etc.); Severe respiratory system diseases (such as bronchial asthma and pulmonary emphysema, etc.).

14.Thrombocytopenic purpura patients; 15.Patients with positive hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) and whose peripheral blood hepatitis B virus (HBV) DNA titer is not within the normal reference range; patients with positive hepatitis C virus (HCV) antibody and whose peripheral blood hepatitis C virus (HCV) RNA is positive; patients with positive human immunodeficiency virus (HIV) antibody; patients with positive cytomegalovirus (CMV) DNA test; patients with positive syphilis test

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-10-21 (Actual); Primary Completion 2028-05-26 (Estimated); Study Completion 2028-05-26 (Estimated)

PRIMARY OUTCOMES:
progression free survial | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No